CLINICAL TRIAL: NCT07250464
Title: Investigation of Motor Evoked Potential and Cortical Silent Period in Migraine Patients
Brief Title: Motor Evoked Potential and Cortical Silent Period in Migraine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IGU-ENF-MK-1
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Migraine; Healty Controls
Keywords: cortical silent period; migraine; single motor unit; transcranial magnetic stimulation
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Magnetic Stimulation; Electromyography

STUDY DESIGN:
Intervention Model Description: Two groups (migraine patients and healthy controls) are evaluated in parallel. Participants and the responsible investigators are blinded to group assignments to reduce bias. Only the staff performing TMS and EMG measurements are aware of group allocation.
Who Masked: Outcomes Assessor
Masking Description: Participants and responsible investigators do not know group assignments. Only the technical staff performing TMS and EMG recordings are aware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraine Patients (Experimental): Adult participants aged 18-45 with a prior diagnosis of migraine according to IHS criteria.
  Transcranial Magnetic Stimulation (TMS)
  Surface Electromyography (sEMG)
  Needle EMG / Single Motor Unit (SMU) Recording
  Interventions: Other: Transcranial Magnetic Stimulation (TMS); Device: Surface Electromyography (sEMG); Other: Needle EMG / Single Motor Unit (SMU) Recording
- Healthy Controls (Sham Comparator): Age- and sex-matched adults without a history of migraine or neurological disorders.
  They undergo the same sEMG and needle EMG/SMU procedures as the migraine group, but the TMS is sham.
  Surface Electromyography (sEMG)
  Needle EMG / Single Motor Unit (SMU) Recording
  Transcranial Magnetic Stimulation (TMS) SHAM
  Interventions: Device: Surface Electromyography (sEMG); Other: Needle EMG / Single Motor Unit (SMU) Recording

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation (TMS) — Non-invasive brain stimulation applied to the primary motor cortex to elicit motor evoked potentials (MEP) and cortical silent periods (CSP).
  70 mm figure-of-eight coil used with Magstim 200² Monophasic Stimulator.
  Arms: Migraine Patients
Device: Surface Electromyography (sEMG) — Bipolar Ag/AgCl electrodes placed over the first dorsal interosseous (FDI) muscle to record muscle responses to TMS.
Other: Needle EMG / Single Motor Unit (SMU) Recording — Sterile Teflon-coated needle electrodes inserted into the FDI muscle to record activity of individual motor units during TMS and voluntary contractions.

SUMMARY:
The primary objective of this study is to assess the level of inhibitory control in the motor cortex of migraine patients using objective and non-invasive methods. To this end, Motor Evoked Potential (MEP) and Cortical Silence Period (CSP) parameters obtained using Transcranial Magnetic Stimulation (TMS) will be measured and comparisons will be made between migraine patients and healthy controls. Since CSP duration is used specifically in the evaluation of GABA-B-mediated inhibitory mechanisms, it has the potential to directly measure the effect of migraine on cortical inhibition.

DETAILED DESCRIPTION:
Rationale and Background:

Migraine is a neurological disorder that significantly impairs individual quality of life and imposes substantial economic burdens on healthcare systems worldwide. Although its pathophysiology is not fully understood, recent research suggests that migraine is associated not only with vascular changes but also with alterations at neurological and cortical levels (Goadsby et al., 2017). Evidence increasingly indicates enhanced excitability and disrupted inhibitory mechanisms in central nervous system regions, including the motor cortex (Coppola et al., 2007).

Transcranial Magnetic Stimulation (TMS) is a non-invasive and reliable neurophysiological technique that stimulates the motor cortex and records muscle responses. Parameters obtained through TMS, such as Motor Evoked Potential (MEP) and Cortical Silent Period (CSP), are used to assess cortical excitability and inhibitory control, respectively (Chen et al., 1999). CSP is particularly useful for evaluating GABA-B-mediated inhibitory mechanisms. The hypothesis that migraine patients exhibit reduced cortical inhibition can be directly tested using CSP measurements.

Previous studies have reported shortened CSP durations and increased MEP amplitudes in migraine patients, suggesting cortical hyperexcitability (Brighina et al., 2002; Afra et al., 1998). However, these findings are inconsistent, and how they vary across migraine subtypes (with aura vs. without aura) remains unclear. Therefore, this study aims to characterize cortical physiological changes in migraine using objective and quantitative measures, filling gaps in the literature and contributing to clinical evaluations. Additionally, the relationship of these parameters with clinical features such as migraine type, duration, and attack frequency will be investigated to lay the groundwork for individualized neurophysiological profiling.

Primary and Secondary Objectives:

Primary Objective:

The primary objective of this study is to objectively evaluate inhibitory control in the motor cortex of migraine patients using non-invasive methods. Motor Evoked Potentials (MEP) and Cortical Silent Periods (CSP) obtained through TMS will be measured and compared between migraine patients and healthy controls. CSP duration, reflecting GABA-B-mediated inhibitory mechanisms, allows direct assessment of migraine's effect on cortical inhibition (Chen et al., 1999).

Secondary Objectives:

Motor Output Analysis: Electromyographic (EMG) signals will be analyzed using Peristimulus Time Histogram (PSTH) and Peristimulus Frequencygram (PSF) methods to assess the temporal pattern and frequency changes of motor unit responses following TMS. PSTH analyzes the timing of individual motor units after stimulation, while PSF provides a more precise view of post-stimulation frequency changes (Türker & Powers, 2001). These analyses help reveal the spinal reflection of cortical stimulation and its effect on motor output.

Biomarker Potential: TMS-derived parameters such as CSP and MEP will be evaluated for their potential as biomarkers of migraine pathophysiology, contributing to the development of objective measures for future diagnosis and treatment.

Expected Benefits:

At the end of this study, it is expected to obtain objective data on motor cortical inhibitory capacity in migraine patients. TMS parameters, particularly CSP and MEP, can be used to understand the neurophysiological basis of migraine. The results may provide:

Improved understanding of cortical excitability and inhibition balance in migraine pathophysiology.

Foundational data for the development of objective diagnostic biomarkers for migraine.

Evidence of cortical dysfunction in migraine patients, supporting personalized treatment approaches.

A comprehensive understanding of motor output from cortical to spinal levels via electrophysiological analyses (PSTH/PSF).

All procedures are non-invasive and safe, providing a reproducible and ethical research approach.

Study Methods:

Participants:

The study will include right-handed individuals aged 18-45 years with a prior diagnosis of migraine according to the International Headache Society (IHS) criteria.

Data Collection:

The study will use non-invasive brain stimulation (TMS) along with surface electromyography (sEMG) and needle EMG. Measurements will be performed both at rest and during voluntary muscle contraction. TMS will be applied over the motor cortex, and muscle responses will be recorded simultaneously using sEMG electrodes. For detailed motor neuron analysis, single motor unit (SMU) recordings will also be obtained.

Needle EMG/SMU Recording:

SMU recordings will use sterile, Teflon-coated needles containing copper wires (approximately 70 μm diameter, 25G) inserted into the first dorsal interosseous (FDI) muscle. Needles will be partially retracted to maintain electrode stability, allowing single motor unit activity to be recorded even during movement.

TMS Application:

TMS will be performed using a Magstim 200^2 Monophasic Stimulator (Magstim Ltd, UK) with a 70 mm figure-of-eight coil placed over the dominant hemisphere's primary motor cortex (M1) corresponding to the FDI muscle. Resting Motor Threshold (RMT) will be determined, followed by stimulation to elicit MEPs.

Surface EMG Recording:

sEMG signals will be obtained using Ag/AgCl electrodes placed over the FDI muscle. Signals will be amplified with a CED 1902 amplifier and digitized via CED 3601 Power 1401 DAC unit. MEP latencies and amplitudes, as well as CSP durations, will be calculated. Participants will maintain ~20% maximal voluntary contraction during measurements.

Data Analysis:

Data will be analyzed using IBM SPSS Statistics 26. Normality will be tested using Kolmogorov-Smirnov and Shapiro-Wilk tests. Parametric data will be analyzed using independent t-tests and ANOVA, while non-parametric data will be analyzed with Mann-Whitney U or Kruskal-Wallis tests. Correlations between clinical parameters (migraine duration, frequency, severity) and neurophysiological measures (MEP, CSP) will be assessed using Pearson or Spearman correlation coefficients, with significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years.
* Right-handed individuals.
* Migraine patients: diagnosed according to International Headache Society (IHS) criteria.
* Healthy controls: no history of migraine or other neurological disorders.
* Able and willing to provide informed consent.

Exclusion Criteria:

* History of epilepsy or other seizure disorders.
* Presence of metal implants, pacemakers, or other contraindications to TMS.
* Pregnancy or breastfeeding.
* History of significant neurological or psychiatric disorders.
* Use of medications that significantly alter cortical excitability (e.g., antiepileptics, benzodiazepines) in the last 2 weeks.
* Any musculoskeletal condition preventing safe participation in EMG/TMS procedures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Cortical Silent Period (CSP) Duration | Single session measurement during TMS
  CSP duration will be recorded from the first dorsal interosseous (FDI) muscle using surface EMG during TMS. CSP reflects GABA-B-mediated cortical inhibitory mechanisms, allowing direct assessment of cortical inhibition in migraine patients compared to healthy controls.

SECONDARY OUTCOMES:
Motor Evoked Potential (MEP) Amplitude | Single session measurement during TMS
  MEP amplitudes will be recorded from FDI muscle using surface EMG. Changes in MEP amplitude reflect cortical excitability and motor output.

OTHER OUTCOMES:
Correlation Between Neurophysiological Parameters and Disease Duration | Single session measurement during TMS
  The relationship between TMS parameters (CSP duration, MEP amplitude) and the duration of the migraine disorder will be assessed using correlation analysis (Pearson or Spearman). Disease duration is determined based on the patient's medical history interview.
Single Motor Unit (SMU) Firing Rate | Single session measurement during TMS
  The discharge rate (firing frequency) of single motor units recorded from the first dorsal interosseous (FDI) muscle using needle EMG during voluntary contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Kemal Sıtkı Türker, Prof. Dr., Principal Investigator — Istanbul Gelisim University, Faculty of Dentistry, Translational Dentistry Research Laboratory
Locations (1):
- Istanbul Gelisim University, Faculty of Dentistry, Translational Dentistry Research Laboratory, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (EMG and TMS measurements) will not be shared outside of the published study results to protect participant confidentiality and privacy.

REFERENCES:
- [Background] Haavik H, Niazi IK, Jochumsen M, Ugincius P, Sebik O, Yilmaz G, Navid MS, Ozyurt MG, Turker KS. Chiropractic spinal manipulation alters TMS induced I-wave excitability and shortens the cortical silent period. J Electromyogr Kinesiol. 2018 Oct;42:24-35. doi: 10.1016/j.jelekin.2018.06.010. Epub 2018 Jun 19. PMID 29936314
- [Background] Ozyurt MG, Haavik H, Nedergaard RW, Topkara B, Senocak BS, Goztepe MB, Niazi IK, Turker KS. Transcranial magnetic stimulation induced early silent period and rebound activity re-examined. PLoS One. 2019 Dec 4;14(12):e0225535. doi: 10.1371/journal.pone.0225535. eCollection 2019. PMID 31800618
- [Background] Todd G, Rogasch NC, Turker KS. Transcranial magnetic stimulation and peristimulus frequencygram. Clin Neurophysiol. 2012 May;123(5):1002-9. doi: 10.1016/j.clinph.2011.09.019. Epub 2011 Oct 22. PMID 22019353
- [Background] Haavik, H., Özyurt, M. G., Niazi, I. K., Nedergaard, R. W., Topkara, B., Yilmaz, G., & Türker, K. S. (2018). Re-investigation on the nature and sign of transcranial magnetic stimulation-induced cortical silent period. In 11th Biennial Meeting of the International Motoneuron Society, IBS, 11-14 June 2018, Boulder, CO, USA (pp. 28-29). Article 46 https://motoneuron2018.org/wp-content/uploads/2018/05/IMS-Poster-Abstracts-2018.pdf
- [Background] Kahya MC, Yavuz SU, Turker KS. Cutaneous silent period in human FDI motor units. Exp Brain Res. 2010 Sep;205(4):455-63. doi: 10.1007/s00221-010-2380-6. Epub 2010 Aug 8. PMID 20694723
- See also: No public protocol page available; contact murkara@gelisim.edu.tr for study information. — https://www.example.com/

DOCUMENTS (2):
  • Study Protocol (2025-10-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT07250464/Prot_000.pdf
  • Informed Consent Form (2025-10-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT07250464/ICF_001.pdf